CLINICAL TRIAL: NCT03002584
Title: International Psychometric Validation Study of the Intestinal Gas Questionnaire (IGQ)
Acronym: PRoVING
Status: Completed | Type: Observational
Sponsor: University Paris 7 - Denis Diderot (Other)
Collaborators: EA 7334, Patient-Centered Outcomes Research (Unknown); University of Manchester (Other); Hospital Vall d'Hebron (Other); Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Olivier CHASSANY, Professor, University Paris 7 - Denis Diderot
Other Study IDs: IGQ
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: IBS - Irritable Bowel Syndrome; General Population
Keywords: IBS, population
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBS & general population: The participants will be given the IGQ questionnaire to complete as well as other self-reported questionnaires.
  Single completion: Participants will have to complete the IGQ, the generic health status EQ-5D questionnaire, the specific FDDQL questionnaire (Functional Digestive Disorders Quality of Life).
  Test-retest: during the second completion within a mean 7-day interval, participants will complete the IGQ and a single global Gastro-Intestinal Well-Being scale.
  Interventions: Other: completion of self-reported questionnaires

INTERVENTIONS:
Other: completion of self-reported questionnaires — Single completion: Participants will have to complete the IGQ, the generic health status EQ-5D questionnaire, the specific FDDQL questionnaire (Functional Digestive Disorders Quality of Life).
  Test-retest: during the second completion within a mean 7-day interval, participants will complete the IGQ and a single global Gastro-Intestinal Well-Being scale

SUMMARY:
Objective: To confirm the psychometrics properties of the Intestinal Gas Questionnaire (IGQ) in subjects with Irritable Bowel Syndrome (IBS) diagnosis and General population both complaining of Gas-Related Symptoms (GRS).

IGQ has been developed previously simultaneously in UK English, French and Spanish through qualitative research with subject interviews. The conceptual framework of the IGQ assesses both GRS and their impact on daily life. Similar concepts were identified for both subjects with IBS diagnosis and general population and complaining of gas-related symptoms.

The IGQ consists of a 24-hour recall symptom diary assessing 7 gas-related symptoms (17 items) and a 7-day recall questionnaire which assesses the impact of those symptoms (26 items)

DETAILED DESCRIPTION:
Observational (non-interventional) study with a cross-sectional part for a subset of adult subjects with a single IGQ completion and a longitudinal cross-over part for a subset of subjects with test-retest IGQ completion for validation of electronic version of IGQ.

300 eligible subjects (100 in each of the 3 countries: France, UK & Spain):

* 180 with IBS diagnosis (60% of recruited subjects)
* 120 from General population (40% of recruited subjects)

ELIGIBILITY:
Inclusion Criteria:

All (subjects with IBS diagnosis and general population):

* Complaining of gas-related symptoms (GRS) of a certain severity level: subjects with IBS diagnosis and general population need to report a score of 4 or greater on at least one symptom on the symptom screening tool
* Cognitive and linguistic capability to complete several self-questionnaires
* BMI > 18.5 and < 30.0 kg/m2
* Agreement of the subject to participate in the study

Subjects with IBS diagnosis:

* IBS diagnosis using Rome III diagnostic criteria for Functional Gastrointestinal Disorders (21)
* IBS severity: IBS-SSS score of 75 to 300

General population:

* Subjects not fulfilling IBS Rome III criteria
* Regular stool frequency (i.e., between 3 and 21 bowel movements per week)

Exclusion criteria

All (subjects with IBS diagnosis and general population):

* Recent (2 last weeks) change in diet or intake of potentially flatulogenic compounds (fiber, lactulose)
* Organic gastrointestinal disease
* Other functional gastrointestinal disorder as defined by Rome III criteria
* Any severe and progressive disease (e.g. depression, cancer, uncontrolled diabetes, rheumatoid arthritis…)
* Any severe psychiatric disorder (e.g. acute episode of schizophrenia or bipolar disorder…)
* Pregnant women
* Being under the direct hierarchy of the investigatorBelonging to the site's staff team

General population:

* Treatment for diarrhea or constipation including lactulose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBS patients and subjects from general population complaining of Gas-Related Symptoms (GRS)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Psychometric validation of the IGQ | cross sectional for 70% of participants and test-retest within an interval of 7 days for 30% of participants
  Stastistical analysis to confirm the psychometric validation of the IGQ questionnaire

SECONDARY OUTCOMES:
Electronic version of the IGQ | During test-retest within an interval of 7 days
  Comparison of scores between paper and electronic version of IGQ

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Chassany, MD, PhD, Study Chair — EA 7334, University Paris-Diderot, Paris; Peter Whorwell, MD, PhD, Principal Investigator — university of Manchester, Manchester; Fernando Azpiroz, MD, PhD, Principal Investigator — Hospital Vall d'Hebron, Barcelona; Benoit Coffin, MD, PhD, Principal Investigator — Hopital Louis Mourier, Colombes; Martin Duracinsky, MD, PhD, Study Director — EA 7334, University Paris-Diderot, Paris
Locations (5):
- Hopital Louis Mourier, Colombes, France
- Spain (3):
  - Centro de salud Chafarinas, Barcelona
  - Horta, Hospital Universitari Vall d'Hebron, Barcelona
  - Centre Mèdic Sant Andreu, Barcelona
- Wythenshawe Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chassany O, Tugaut B, Marrel A, Guyonnet D, Arbuckle R, Duracinsky M, Whorwell PJ, Azpiroz F. The Intestinal Gas Questionnaire: development of a new instrument for measuring gas-related symptoms and their impact on daily life. Neurogastroenterol Motil. 2015 Jun;27(6):885-98. doi: 10.1111/nmo.12565. Epub 2015 Apr 6. PMID 25846412
- See also: Results of the qualitative analysis — http://onlinelibrary.wiley.com/doi/10.1111/nmo.12565/abstract